CLINICAL TRIAL: NCT02687256
Title: Evaluation of Extended Infusion Set Wear Using the Medtronic Extended Wear Sof-set Infusion Set
Brief Title: Evaluation of Extended Infusion Set Wear Using Medtronic Extended Wear Sof-set Infusion Set
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Bruce A. Buckingham, M.D., Stanford University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 36142
Record Dates: First submitted 2016-02-09; First posted 2016-02-22 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Heparin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (9):
- Protocol 1: Standard then Extended Set (Experimental): Participants will wear the control (standard) infusion set for 1 week, then switch to the experimental Extended Wear infusion set in combination with Heparin 400 IU for 1 week, then will repeat the cycle for a total of 4 weeks.
  Interventions: Device: Extended Wear infusion set; Device: Standard Infusion set; Drug: Heparin
- Protocol 1: Extended then Standard Set (Experimental): Participants will wear the experimental Extended Wear infusion set in combination with Heparin 400 IU for 1 week, then switch to the control (standard) infusion set for 1 week, then will repeat the cycle for a total of 4 weeks.
  Interventions: Device: Extended Wear infusion set; Device: Standard Infusion set; Drug: Heparin
- Protocol 2 (Part 1): Sequence 1 (Experimental): Participants will wear the control (standard) infusion set for 1 week, then the Extended Wear infusion set with heparin at 40 IU (week 1), 80 IU (week 2), 120 IU (week 3), and 200 IU (week 4).
  Interventions: Device: Extended Wear infusion set; Device: Standard Infusion set; Drug: Heparin
- Protocol 2 (Part 1): Sequence 2 (Experimental): Participants will wear the Extended Wear infusion set with heparin at 40 IU (week 1), 80 IU (week 2), 120 IU (week 3), and 200 IU (week 4), then the control (standard) infusion set (week 5).
  Interventions: Device: Extended Wear infusion set; Device: Standard Infusion set; Drug: Heparin
- Protocol 2 (Part 1): Sequence 3 (Experimental): Participants will wear the Extended Wear infusion set with heparin at 80 IU (week 1), 120 IU (week 2), and 200 IU (week 3), then the control (standard) infusion set (week 4), then the Extended Wear infusion set with heparin at 40 IU (week 5).
  Interventions: Device: Extended Wear infusion set; Device: Standard Infusion set; Drug: Heparin
- Protocol 2 (Part 1): Sequence 4 (Experimental): Participants will wear the Extended Wear infusion set with heparin at 120 IU (week 1), and 200 IU (week 2), then the control (standard) infusion set (week 3), then the Extended Wear infusion set with heparin at 40 IU (week 4), and 80 IU (week 5).
  Interventions: Device: Extended Wear infusion set; Device: Standard Infusion set; Drug: Heparin
- Protocol 2 (Part 1): Sequence 5 (Experimental): Participants will wear the Extended Wear infusion set with heparin at 200 IU (week 1), then the control (standard) infusion set (week 2), then the Extended Wear infusion set with heparin at 40 IU (week 3), 80 IU (week 4), and 80 IU (week 5).
  Interventions: Device: Extended Wear infusion set; Device: Standard Infusion set; Drug: Heparin
- Protocol 2 (Part 2): Standard then Extended Set (Experimental): Participants will wear the control (standard) infusion set for 1 week, then switch to the experimental Extended Wear infusion set in combination with Heparin 80 IU for 1 week, then will repeat the cycle for a total of 4 weeks.
  Interventions: Device: Extended Wear infusion set; Device: Standard Infusion set; Drug: Heparin
- Protocol 2 (Part 1): Extended then Standard Set (Experimental): Participants will wear the experimental Extended Wear infusion set in combination with Heparin 80 IU for 1 week, then switch to the control (standard) infusion set for 1 week, then will repeat the cycle for a total of 4 weeks.
  Interventions: Device: Extended Wear infusion set; Device: Standard Infusion set; Drug: Heparin

INTERVENTIONS:
Device: Extended Wear infusion set — For two of the 4 weeks the Extended Wear insulin infusion set will be used.
Device: Standard Infusion set — For two of the 4 weeks the Standard infusion set will be used
  Other Names: Minimed
Drug: Heparin

SUMMARY:
This is a blinded cross-over study to see if extended wear insulin infusion sets can prolong insulin infusion set wear up to 7 days in adults with Type 1 Diabetes.

DETAILED DESCRIPTION:
This is a double blinded cross-over study. Subjects will be asked to wear infusion set either a standard infusion set or an extended wear infusion set. They will wear each infusion set twice, and the order of infusion set wear will be randomized with the first infusion set wear and then alternated over 4 weeks. By performing a cross over study using both experimental infusion sets and standard infusion sets, the investigators hope to see whether there is a benefit to using an extended wear infusion set.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes for at least one year and using an insulin pump for at least 12 months
2. The diagnosis of type 1 diabetes is based on the investigator's judgment; C-peptide level and antibody determinations are not needed.
3. Age 18 to 55 years
4. Hemoglobin A1c level less than or equal to 8.5%
5. Willing to use Novolog insulin while they are participating in the study
6. Total daily insulin dose is at least 0.3 units/kg/day
7. For females, not currently known to be pregnant
8. An understanding of and willingness to follow the protocol and sign the informed consent
9. Willingness to wear the experimental insulin infusion sets throughout the study
10. Must be able to understand spoken and written English

Exclusion Criteria:

1. Diabetic ketoacidosis in the past 3 months
2. blood urea nitrogen (BUN), Creatinine, or liver function test (ALT or AST) more than three times the upper limit of normal, or thrombocytopenia
3. Severe hypoglycemia resulting in seizure or loss of consciousness in the 3 months prior to enrollment
4. Pregnant or lactating females
5. Known tape allergies
6. Current treatment for a seizure disorder
7. Cystic fibrosis
8. Active infection
9. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:
10. Inpatient psychiatric treatment in the past 6 months for either the subject or the subject's primary care giver (i.e., parent or guardian)
11. Presence of a known adrenal disorder
12. If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study
13. Abuse of alcohol
14. Dialysis for renal failure

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Time to an infusion set failure due to an occlusion | within 1 week
  Glucose >250 mg/dL with failure of a correction dose to lower the glucose by 50 mg/dL, or ketones > or = 0.6 mg/dL with a glucose reading of >250 mg/dL (in the absence of illness), or a pump occlusion alarm

SECONDARY OUTCOMES:
signs of infection at insulin infusion site | 1 week
  erythema or induration of > 1cm in diameter at injection site

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Buckingham, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
To maintain the integrity of this research study, the subject is told they may not have access to any health information developed as part of this study until it is completed.